CLINICAL TRIAL: NCT07403084
Title: Post-market Clinical Follow-up Study of NEMOST V2 Growing Domino
Brief Title: Post-market Clinical Follow-up Study of NEMOST V2
Acronym: NEMOST V2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EUROS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-304-02
Record Dates: First submitted 2026-01-28; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Scoliosis Neuromuscular; Scoliosis Idiopathic; Consent Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NEMOST V2 (Experimental)
  Interventions: Device: NEMOST V2 growing domino

INTERVENTIONS:
Device: NEMOST V2 growing domino — The NEMOST spinal implant is a growth domino intended for the surgical treatment of progressive scoliosis in children.

SUMMARY:
The NEMOST spinal implant is a growth domino intended for the surgical treatment of progressive scoliosis in children.

As part of post-market surveillance, EUROS is conducting a retrospective and prospective study to collect clinical and radiological data on the NEMOST growth domino.

Retrospective and prospective multicenter post-market surveillance clinical study.

This study is interventional, non-randomized, and uncontrolled. The primary objective of this clinical study is to monitor complications related to the NEMOST growth domino during a 5-year postoperative follow-up in patients treated for progressive scoliosis in children.

The secondary objective of this clinical study is to monitor the performance of the NEMOST growth domino during a 5-year postoperative follow-up in patients treated for progressive scoliosis in children.

The study will include 140 patients.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic, congenital, neuromuscular, or syndromic scoliosis : Progressive spinal deformity not managed by orthopedic treatment, and requiring primary surgical intervention.
* The patient, as well as their parents or legal guardians, are informed of the participation in the study.
* Patients aged from 5 to 17 yeas old, excepted the one who still have a potential for growth

Exclusion Criteria:

* signs of local inflammation;
* acute or chronic, local or systemic infections ;
* non-reducible scoliosis ;
* pathological obesity ;
* allergy or intolerance to implanted materials;
* insufficiency or absence of tissue coverage. The NEMOST implant should not be used in a spine that has already been instrumented or fused.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2033-12-19 (Estimated); Study Completion 2033-12-19 (Estimated)

PRIMARY OUTCOMES:
Complication rate | 5 years
  The safety of the device will be studied by monitoring all complications, reinterventions and revisions.

SECONDARY OUTCOMES:
Cobb angle (°) | 5 years
  Comparison between preoperative measures, immediate postoperative measures and each visit measures.
  Measured on seated or standing anteroposterior and lateral X-ray images by identifying the most tilted vertebrae at the top and bottom of the spinal curve, drawing lines along their endplates, and calculating the angle formed by the intersection of perpendiculars to these lines. Normal value for Cobb angle is <10° for no or benign scoliosis, medium scoliosis is defined between 15 and 35°, important scoliosis is defined as between 35 and 60° and very important scoliosis corresponds to angle > 65°. The Cobb angle correction, used to compare pre and postoperative angle is defined as 100*(preoperative value - postoperative value) / postoperative value.
Early-Onset Scoliosis questionnaire 24 items (EOSQ-24) | 5 years
  Considering clinical evaluation, the EOSQ-24 auto questionnaire addressed to patients' parents was selected. The 24-Item Early-onset Scoliosis Questionnaire (EOSQ-24) is a locally validated measurement tool to evaluate the overall impact of early onset scoliosis on patients' physical, psychological, and socio-economic well-being. Clinical results are assessed thanks to the EOSQ-24 quality of life questionnaire. It is divided in 11 themes, for which a score is calculated over 100. Each item is composed of 1 to 5 questions rated from 1 to 5, 5 being the best score. These scores will be between 0 to 100.
  Comparison between preoperative measures, immediate postoperative measures and each visit measures.
Pelvic obliquity (°) | 5 years
  Measured on seated or standing anteroposterior and lateral X-ray images by drawing a line between the iliac crests (or the inferior aspects of the sacroiliac joints) and calculating the angle between this line and a horizontal reference line. Normal value is 0°.
  Comparison between preoperative measures, immediate postoperative measures and each visit measures.
Thoracic kyphosis (°) | 5 years
  Measured on seated or standing anteroposterior and lateral X-ray images by calculating the Cobb angle between the superior endplate of the upper thoracic vertebra and the inferior endplate of the lower thoracic vertebra defining the kyphotic curve (commonly T4-T12).
  Comparison between preoperative measures, immediate postoperative measures and each visit measures.
Lumbar lordosis (°) | 5 years
  Measured on seated or standing anteroposterior and lateral X-ray images by calculating the Cobb angle between the superior endplate of the upper lumbar vertebra and the superior endplate of the sacrum (commonly L1-S1).
  Comparison between preoperative measures, immediate postoperative measures and each visit measures.
  Normal value ranges from 20 to 60°.
T1-T12 and T1-S1 length (mm) | 5 years
  T1-T12 length is measured on a standing or seated anteroposterior spinal radiograph as the linear distance between the midpoint of the superior endplate of T1 and the midpoint of the inferior endplate of T12.
  T1-S1 length is measured on a standing or seated anteroposterior spinal radiograph as the linear distance between the midpoint of the superior endplate of T1 and the midpoint of the superior endplate of S1.
  Comparison between preoperative measures, immediate postoperative measures and each visit measures.
Respiratory functional exploration | 5 years
  Pulmonary function testing is performed in a seated or supine position by measuring Total Lung Capacity (TLC, mL) and Vital Capacity (VC, mL) using standardized pulmonary function tests.
  Comparison between preoperative measures and each visit measures.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Solla, MD, Principal Investigator — CHU NICE
Locations (5):
- France (5):
  - Hopital Lenval Nice, Nice, Provence-Alpes-Côte d'Azur Region
  - CHU Pellegrin, Bordeaux
  - Hospices Civils de Lyon, Lyon
  - Hopital Armand Trousseau, Paris
  - Hopital Necker, Paris

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-12-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT07403084/Prot_SAP_ICF_000.pdf